CLINICAL TRIAL: NCT04276285
Title: Impact of Laparoscopic Versus Ultrasound-Guided Subcostal Transversus Abdominis Plane Block on Pain and Recovery After Laparoscopic Cholecystectomy: A Randomized Double-Blinded Controlled Study
Brief Title: Laparoscopic Versus US-Guided Subcostal TAP Block After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mansoura124
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Cholecystitis; Gallstone
MeSH Terms: conditions — Cholecystitis; Gallstones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic TAP (Active Comparator): Subcostal TAP block will be performed after surgery under laparoscopic guidance
  Interventions: Procedure: Laparoscopic TAP
- US TAP (Active Comparator): Subcostal TAP block will be performed after surgery under ultrasound guidance
  Interventions: Procedure: US TAP
- No TAP (No Intervention): No TAP block will be performed

INTERVENTIONS:
Procedure: Laparoscopic TAP — Subcostal TAP block will be performed after surgery under laparoscopic guidance
  Arms: Laparoscopic TAP
Procedure: US TAP — Subcostal TAP block will be performed after surgery under US guidance
  Arms: US TAP

SUMMARY:
Zaghiyan et al hypothesized that Laparoscopic TAP was noninferior to US-TAP and performed a randomized clinical trial comparing Laparoscopic TAP, US-TAP, and no TAP in minimally invasive colorectal surgery. The authors reported that LTAP was superior to UTAP in achieving pain control and minimizing opioid use in the first 24 hours after colorectal surgery.

This prospective randomized, controlled trial will be performed to assessed the efficacy of laparoscopic subcostal TAP block (LSTAP) compared to ultrasound-guided subcostal TAP (USTAP) block after laparoscopic cholecystectomy regarding postoperative pain scores in the first 24-hours after the intervention and analgesic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients of either gender who will undergo laparoscopic cholecystectomy will be recruited to the study.

Exclusion Criteria:

* Pregnant women
* Patients who will undergo open cholecystectomy
* Patients who will need conversion to conventional open cholecystectomy
* Patients with ASA III classification or higher
* Patients who will undergo laparoscopic cholecystectomy together with other abdominal interventions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 24 hours after cholecystectomy
  pain will be assessed with visual analogue scale from 0-10

SECONDARY OUTCOMES:
Analgesic requirement | 24 hours after cholecystectomy
  the need for intravenous analgesia after surgery calculated as the cumulative dose of analgesic administered over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No